CLINICAL TRIAL: NCT03583060
Title: Interoceptive Engagement in Response to Mindful Awareness in Body-oriented Therapy: A Pilot Test Comparison
Brief Title: Interoceptive Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Cynthia Price, Research Assoc. Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00003441
Record Dates: First submitted 2018-06-26; First posted 2018-07-11 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MABT (Experimental): Receive 8 weekly sessions of Mindful Awareness in Body-oriented Therapy (MABT).
  Interventions: Behavioral: Mindful Awareness in body-oriented therapy
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Mindful Awareness in body-oriented therapy — teaches interoceptive awareness skills for self care
  Arms: MABT

SUMMARY:
The proposed project is the first pilot test to examine interoceptive function as a mechanistic biomarker underlying Mindful Awareness in Body-oriented Therapy (MABT). MABT, an empirically-validated and manualized protocol is explicitly designed to teach interoceptive awareness skills for emotion regulation and is thus an ideal intervention approach in which to address this gap in research. This study uses a two group, randomized design to examine neural and physiological biomarkers in response to MABT. Twenty-four individuals reporting moderate stress will be recruited from the community and randomized to 8-week MABT intervention or the control condition. The study aims are to: 1) evaluate whether interoceptive training improves interoceptive function in the MABT vs control condition, and 2) explore whether changes in interoceptive function correlate with improved health outcomes. Analyses will include within and between-group ANOVA of brain activity with symptom change as a covariate. This is the first study to test whether a clinical intervention aimed specifically at cultivating interoceptive awareness effects change on interoceptive biomarkers. The results will support larger NIH proposals to more comprehensively validate neuro and behavioral biomarkers of interoceptive training to enhance mental health, particularly targeting depression and substance use disorder that have identified interoceptive dysfunction and poor emotion regulation.

ELIGIBILITY:
Inclusion Criteria:

* adult (over 18)
* Perceived Stress Scale scores indicating moderate stress levels
* naive to mindfulness-based approaches (no prior experience)
* agrees to forgo (non-study) manual therapies (e.g., massage) and mind-body therapies (e.g., mindfulness meditation) for 3 months (baseline to post-test)
* fluent in English
* can attend MABT and assessment sessions
* right-handed (for uniformity of neuroimaging results)

Exclusion Criteria:

* lifetime diagnosis of mental health disorder
* unable to complete study participation (includes planned relocation, pending inpatient treatment, planned extensive surgical procedures, etc.)
* cognitive impairment, assessed by the Mini-Mental Status Exam (MMSE) if demonstrated difficulty comprehending the consent
* use of medications in the past 30 days that affect hemodynamic response
* lifetime head injuries or loss of consciousness longer than 5 min
* currently pregnant
* contraindications for MRI, e.g., claustrophobia, metal objects in body, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
interoceptive function | 10 weeks
  Functional magnetic resonance imaging (fMRI)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Price, PhD, Principal Investigator — University of Washington; Norman Farb, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No